CLINICAL TRIAL: NCT02060305
Title: A Pilot Study About the Safety and Efficacy of Intra-articular Bevacizumab (Avastin) for Recurrent Hemarthroses at Target Joints With Chronic Hemophilic Synovitis
Brief Title: Intra-articular Bevacizumab for Recurrent Hemarthroses at Target Joints With Chronic Hemophilic Synovitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Very slow enrollment
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, Statistical Center, NTUHCTC, National Taiwan University Hospital, National Taiwan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201305041MINB
Record Dates: First submitted 2014-02-05; First posted 2014-02-12 (Estimated); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Hemophilia; Synovitis
MeSH Terms: conditions — Hemophilia A; Synovitis | interventions — Bevacizumab; Injections, Intra-Articular

STUDY DESIGN:
Intervention Model Description: Open-label
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab (Experimental): Bevacizumab intra-articular injection; dose 20mg~40mg every 28 days for 4 times
  Interventions: Drug: Bevacizumab intra-articular injection

INTERVENTIONS:
Drug: Bevacizumab intra-articular injection — Bevacizumab, 20~40mg, intra-articular injection every 28 days for 4 times
  Other Names: Bevacizumab (Avastin) intra-articular injection

SUMMARY:
Primary Objective The efficacy of intra-articular bevacizumab injection for secondary prevention of recurrent hemarthroses for hemophilia patients who has had target joints with chronic synovitis. The safety profiles of intra-articular bevacizumab injection for hemophilia patients.

Study Population Adult hemophilia patients who have had one or more target joints with chronic synovitis and recurrent hemarthroses.

Investigational therapy: Intra-articular injection of Bevacizumab (20 or 40 mg/ 0.8 or 1.6 ml/ dose) every month (28 days) for up to 4 months, depending on the improvement of target joint bleeding.

Study Design The estimated study period is between Jan 2014 and Dec 2015. Totally 10 joints will be enrolled for this pilot study. Before enrollment, the joint(s) will be evaluated for their severity both clinically (by 10-point Pain Score, range of motion for the target joint, and World Federation of Hemophilia Score) and by MRI (using the compatible MRI scales developed by International Prophylaxis Study Group [IPSG]). Intra-articular injection of bevacizumab will be administered, after prophylactic factor supplementation, every month for up to four injections. In the first four patients, 20mg of bevacizumab will be administered. If there are no Gr 3 or Gr4 dose-limiting toxicities, bevacizumab dose will be escalated to 40mg in the other 6 patients. Before every procedure, the plasma and the synovial fluid samples will be collected for VEGF quantification for the correlative biomarker study. After completing the protocol treatment, the efficacy parameters as well as the safety profiles will be evaluated.

DETAILED DESCRIPTION:
Hypothesis: The mechanism of recurrent hemarthroses (joint bleeds) resulted from chronic synovitis of target joints in hemophilic patients is thought to be a VEGF-based neo-angiogenic process. Local anti-VEGF therapy with intra-articular bevacizumab (Avastin), a VEGF-neutralizing monoclonal antibody that can efficiently antagonize VEGF activity, may block the process and decrease the frequency of recurrent bleeding episodes. In addition, we proved that intra-articular injection of bevacizumab in rat model is safe without significant local or systemic adverse events.

Primary Objective The efficacy of intra-articular bevacizumab injection for secondary prevention of recurrent hemarthroses for hemophilia patients who has had target joints with chronic synovitis. The safety profiles of intra-articular bevacizumab injection for hemophilia patients.

Study Population Adult hemophilia patients who have had one or more target joints with chronic synovitis and recurrent hemarthroses.

Investigational therapy: Intra-articular injection of Bevacizumab (20 or 40 mg/ 0.8 or 1.6 ml/ dose) every month (28 days) for up to 4 months, depending on the improvement of target joint bleeding.

Study Design The estimated study period is between Jan 2014 and Dec 2015. Totally 10 joints will be enrolled for this pilot study. Before enrollment, the joint(s) will be evaluated for their severity both clinically (by 10-point Pain Score, range of motion for the target joint, and World Federation of Hemophilia Score) and by MRI (using the compatible MRI scales developed by International Prophylaxis Study Group [IPSG]). Intra-articular injection of bevacizumab will be administered, after prophylactic factor supplementation, every month for up to four injections. In the first four patients, 20mg of bevacizumab will be administered. If there are no Gr 3 or Gr4 dose-limiting toxicities, bevacizumab dose will be escalated to 40mg in the other 6 patients. Before every procedure, the plasma and the synovial fluid samples will be collected for VEGF quantification for the correlative biomarker study. After completing the protocol treatment, the efficacy parameters as well as the safety profiles will be evaluated.

Assessments The efficacy: the differences of total episodes of recurrent hemarthroses within 3 months before and after completing bevacizumab intra-articular injection. Post-procedure target joints bleedings will be recorded at intervals of 1st, 3rd, 6th, and 12th months. The total absence of haemarthrosis (zero bleeding) is rated as "excellent" response; bleeding reduction between 75% and 99% is rated "good", between 50% and 74% as "fair", and below 50% as "poor".

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older, with a diagnosis of hemophilia A or B.
2. Subjects with target one or more target joints of chronic synovitis with recurrent hemarthroses more than 2 times in recent 6 months. The target joint(s) are limited to knee, elbow, or ankle, with substantial severity (World Federation of Hemophilia Score =2~3)
3. White cell count ≧ 3000/μL, Hemoglobin level ≧ 10 g/dL, and platelets ≧ 100,000/μL
4. Serum creatinine ≦1.5 X the upper limit of normal (ULN)
5. Total bilirubin ≦1.5 X ULN; aspartate and alanine aminotransferase (AST, ALT) ≦2.0 x ULN.
6. Willingness and ability to comply with the study scheduled visits, treatment plans, laboratory tests, and other procedures, including the completion of patient questionnaires.
7. Women of childbearing potential must have a negative serum pregnancy test done 1 week prior to the administration of the study drug. She and her partner should prevent pregnancy (oral contraceptives, intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly or surgically sterile) up to at least 6 months after last treatment completion or the last drug dose, whatever happens first.
8. Eastern Cooperative Oncology Group (ECOG) performance status: 0~2
9. Signed written informed consent according to ICH/GCP and the local regulations (approved by the Institutional Review Board [IRB]/Independent Ethics Committee [IEC]) will be obtained prior to any study specific screening procedures.

Exclusion Criteria:

1. Subjects with known HIV infection.
2. Subjects whose target joints have been heavily damaged into deformity or arthropathy, or whose target joints cannot receive intra-articular injection.
3. Subjects who cannot receive MRI study.
4. Subjects with uncontrolled hypertension (systolic blood pressure > 160 mm Hg, diastolic blood pressure > 90 mm Hg).
5. Subjects who experienced major surgical procedures, open biopsy or significant traumatic injury within 28 days prior to the first dose of Bevacizumab administration (Patients must have recovered from any major surgery), or who have anticipation of need for major surgical procedures during the course of the study.
6. Subjects with serious non-healing wound or ulcer.
7. Subjects with clinically significant (i.e. active) cardiovascular disease. For example, cerebrovascular accidents or stroke in the preceding six months, myocardial infarction or unstable angina in the preceding six months, New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication.
8. Pregnancy (positive serum pregnancy test) and lactation
9. Subjects who have other impaired major organ dysfunction, active infection, abnormal laboratory or physical findings, or co-morbidities that, in the investigators' adjustment, may substantially increase the risk associated with the patients' participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-02-01; Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Recurrent hemarthroses rate | one year
  The efficacy of intra-articular bevacizumab injection for secondary prevention of recurrent hemarthroses for hemophilia patients who has had target joints with chronic synovitis. The efficacy will be measure by the recurrent hemarthroses rate after the investigational therapy

SECONDARY OUTCOMES:
The dynamics of serum and synovial fluid VEGF concentrations | one year
The vasculature changes by MR image study | one year
The pain score during the intra-articular injection procedure | 6 months
The frequency and severity of adverse effects during the study period | one year
  The adverse effects, both systemic (Ex. hypertension, proteinuria, or bleeding episodes), and localized (Ex. joint internal bleeding or local symptoms), will be monitored and recorded during the investigation period.

CONTACTS AND LOCATIONS:
Overall Officials: Shang-Ju Wu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Hematology Division, National Taiwan University Hospital, Taipei, Taiwan